CLINICAL TRIAL: NCT01749904
Title: A Randomized, Multicenter, Double-Masked, Parallel-Group Study Comparing the Safety and Efficacy of BOL-303259-X Ophthalmic Solution With Timolol Maleate Ophthalmic Solution 0.5% in Subjects With Open-Angle Glaucoma or Ocular Hypertension.
Brief Title: Comparing Safety and Efficacy of BOL-303259-X With Timolol Maleate in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Acronym: APOLLO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 769
Record Dates: First submitted 2012-12-11; First posted 2012-12-17 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-08

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — BOL 303259-X; Timolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BOL-303259-X (Experimental): BOL-303259-X ophthalmic solution QD (PM) and vehicle QD (AM) administered for 3 months (Visit 6) into the study eye(s).
  Interventions: Drug: BOL-303259-X
- Timolol (Active Comparator): Timolol maleate ophthalmic solution, 0.5%, administered BID for 3 months (Visit 6) into study eye(s).
  Interventions: Drug: Timolol; Drug: BOL-303259-X

INTERVENTIONS:
Drug: BOL-303259-X — Topical ocular BOL-303259-X will be administered QD in the evening and its vehicle administered QD in the morning for 3 months (visit 6).
  Arms: BOL-303259-X
Drug: Timolol — Timolol will be administered BID once in the morning and once in the evening for 3 months (Visit 6)
  Arms: Timolol
Drug: BOL-303259-X — All participants will receive topical ocular BOL-303259-X QD in the evening for an additional 9 months from Visit 6 through Visit 9 (1 year)

SUMMARY:
In participants with a diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT), the primary objective is to demonstrate that the mean IOP reduction after 3 months of treatment with BOL-303259-X once daily (QD) is non-inferior to timolol maleate 0.5% twice daily (BID). The secondary objective is to demonstrate the superiority of BOL-303259-X QD to timolol maleate 0.5% BID. This assessment will be performed if the non-inferiority of BOL-303259-X QD to timolol maleate 0.5% BID is determined. An open label safety phase will be conducted at the end of Visit 6 (3 months) where all participants will receive BOL-303259-X QD for an additional 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of OAG (including pigmentary or pseudoexfoliative) or OHT in 1 or both eyes.
* Participants must meet the following IOP requirements at Visit 3
* mean/median IOP ≥ 24 mmHg at a minimum of 2 time points in the same eye
* IOP ≤ 36 mmHg at all 3 measurement time points in both eyes.
* Participants with a best-corrected visual acuity (BCVA), using the Early Treatment of Diabetic Retinopathy Study (ETDRS) protocol, of +0.7 logMAR units (Snellen equivalent of approximately 20/100) or better in either eye.

Exclusion Criteria:

* Participants with known hypersensitivity or contraindications to latanoprost, NO treatment, timolol maleate, other beta-adrenergic receptor antagonists or any of the ingredients in the study drugs.
* Participants with a central corneal thickness greater than 600 μm in either eye.
* Participants with advanced glaucoma and participants with a cup/disc ratio greater than 0.8 or a history of split fixation, or a field loss threatening fixation in either eye.
* Participants who do not have an intact posterior capsule in either eye .
* Participants with aphakia in either eye.
* Participants with previous or active corneal disease in either eye.
* Participants with current or a history of severe dry eye in either eye.
* Participants with current or a history of optic disc hemorrhage in either eye.
* Participants with current or a history of central/branch retinal vein or artery occlusion in either eye.
* Participants with current or a history of macular edema in either eye.
* Participants with very narrow angles (3 quadrants with less than Grade 2 according to Shaffer's anterior chamber angle grading system) and Participants with angle closure,congenital, and secondary glaucoma, and participants with history of angle closure in either eye.
* Participants with a diagnosis of a clinically significant or progressive retinal disease in either eye.
* Participants with any intraocular infection or inflammation in either eye within 3 months(90 days) prior to Visit 1 (Screening).
* Participants with a history of ocular laser surgery in either eye within the 3 months(90 days) prior to Visit 1 (Screening).
* Participants with a history of incisional ocular surgery or severe trauma in either eye within 3 months (90 days) prior to Visit 1 (Screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2015-06-02 (Actual); Study Completion 2015-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Vittitow, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Inc., Rochester, New York, United States

REFERENCES:
- [Result] Weinreb RN, Scassellati Sforzolini B, Vittitow J, Liebmann J. Latanoprostene Bunod 0.024% versus Timolol Maleate 0.5% in Subjects with Open-Angle Glaucoma or Ocular Hypertension: The APOLLO Study. Ophthalmology. 2016 May;123(5):965-73. doi: 10.1016/j.ophtha.2016.01.019. Epub 2016 Feb 11. PMID 26875002
- [Result] Weinreb RN, Liebmann JM, Martin KR, Kaufman PL, Vittitow JL. Latanoprostene Bunod 0.024% in Subjects With Open-angle Glaucoma or Ocular Hypertension: Pooled Phase 3 Study Findings. J Glaucoma. 2018 Jan;27(1):7-15. doi: 10.1097/IJG.0000000000000831. PMID 29194198

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BOL-303259-X | Timolol
Started | 286 (randomized population) | 134 (randomized population)
Completed | 264 (randomized population) | 123 (randomized population)
Not Completed | 22 | 11

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population. Of the 420 subjects randomized, 418 instilled at least one dose of study medication and were included in the safety population, whereas one subject did not have any post-baseline efficacy reading, hence 417 subjects were included in the Intent-to-treat population
Groups:
- BOL-303259-X: BOL-303259-X ophthalmic solution QD (PM) and vehicle QD (AM) administered for 3 months (Visit 6) into the study eye during the efficacy phase, and for an additional 9 months from Visit 6 through Visit 9 (1 year) during the open label safety extension phase
- Timolol: Timolol maleate ophthalmic solution, 0.5%, administered BID for 3 months (Visit 6) into study eye. thereafter these subjects were switched to receive topical ocular BOL-303259-X QD in the evening for an additional 9 months from Visit 6 through Visit 9 (1 year)
- Total: Total of all reporting groups
Arm/Group | BOL-303259-X | Timolol | Total
Number analyzed (Participants) | 284 | 133 | 417
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (10.32) | 63.1 (11.23) | 64.2 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 77 | 243
  Male | 118 | 56 | 174
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 13 | 43
  Not Hispanic or Latino | 254 | 120 | 374
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 64 | 24 | 88
  White | 217 | 108 | 325
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean IOP
Description: Mean intraocular pressure (IOP) in study eye measured at the specified time points: 8 AM, 12 PM, and 4 PM at Visit 4(Week 2), Visit 5 (Week 6), and Visit 6 (Month 3).
Time Frame: 8 AM, 12 PM, and 4 PM at Visit 4(Week 2), Visit 5 (Week 6), and Visit 6 (Month 3)
Population: Intent-to-treat population with LOCF
Measure: Least Squares Mean (Standard Deviation); unit: mm Hg
Arm/Group | BOL-303259-X | Timolol
Number analyzed (Participants) | 284 | 133
mm Hg
  8 am week 2: number analyzed (Participants) | 282 | 133
  8 am week 2 | 18.61 (3.544) | 19.84 (3.651)
  12 pm week 2: number analyzed (Participants) | 282 | 131
  12 pm week 2 | 18.00 (3.376) | 19.37 (3.696)
  4 pm week 2: number analyzed (Participants) | 281 | 131
  4 pm week 2 | 18.09 (3.293) | 19.20 (3.359)
  8 am week 6: number analyzed (Participants) | 283 | 133
  8 am week 6 | 18.59 (3.525) | 19.63 (3.243)
  12 pm week 6: number analyzed (Participants) | 283 | 131
  12 pm week 6 | 17.84 (3.305) | 19.09 (3.230)
  4 pm week 6: number analyzed (Participants) | 284 | 131
  4 pm week 6 | 17.82 (3.513) | 19.09 (3.492)
  8 am Month 3: number analyzed (Participants) | 283 | 133
  8 am Month 3 | 18.71 (3.382) | 19.73 (2.230)
  12 pm Month 3: number analyzed (Participants) | 283 | 131
  12 pm Month 3 | 17.88 (3.409) | 19.15 (3.311)
  4 pm Month 3: number analyzed (Participants) | 284 | 131
  4 pm Month 3 | 17.83 (3.521) | 19.15 (3.643)
Statistical Analysis 1: Comparison: BOL-303259-X vs Timolol; Test type: Non-Inferiority — The 2 treatments were compared for each time point by visit. LS mean of each treatment group, the difference in the LS mean, and the 2-sided 95% CI for the difference were obtained. Noninferiority could be claimed if the upper limit of the CIs <1.5 mmHg at all time points of each visit and <1.00 mmHg for at least 5 out of the 9 time points. If noninferiority was determined, superiority at each time point could be claimed if the upper limit of the 95% CI<0 mmHg at all time points of each visit; p < 0.01, ANCOVA — The ANCOVA results for the comparison of LS means of mean IOP between treatment groups demonstrated noninferiority of BOL-303259-X to timolol and also superiority of BOL-303259-X to timolol

2. Secondary Outcome: Response Rate - IOP ≤ 18 mm Hg
Description: Percentage of participants with IOP ≤ 18 mm Hg consistently at all 9 time points in the first 3 months
Time Frame: 8 AM, 12 PM, and 4 PM at Visit 4(Week 2), Visit 5 (Week 6), and Visit 6 (Month 3).
Population: Intent-to-treat population with LOCF
Measure: Count of Participants; unit: Participants
Arm/Group | BOL-303259-X | Timolol
Number analyzed (Participants) | 284 | 133
Participants | 65 | 15
Statistical Analysis 1: Comparison: BOL-303259-X vs Timolol; Test type: Other; p = 0.005, Chi-squared

3. Secondary Outcome: Response Rate - IOP Reduction ≥ 25%
Description: Percentage of participants with IOP reduction ≥ 25% consistently at all 9 time points in the first 3 months
Time Frame: 8 AM, 12 PM, and 4 PM at Visit 4(Week 2), Visit 5 (Week 6), and Visit 6 (Month 3).
Population: Intent-to-treat with LOCF
Measure: Count of Participants; unit: Participants
Arm/Group | BOL-303259-X | Timolol
Number analyzed (Participants) | 284 | 133
Participants | 99 | 26
Statistical Analysis 1: Comparison: BOL-303259-X vs Timolol; Test type: Other; p = 0.001, Chi-squared

4. Other Pre Specified Outcome: Number of Participants With Ocular and Systemic Adverse Events
Description: Following assessments through Visit 6 (Month 3), all participants, irrespective of previous randomization, converted to a single open label safety arm receiving BOL-303259-X QD in the evening. Adverse events were recorded throughout the comparative efficacy phase and open label extension phase.
Time Frame: 12 months
Population: Safety population (analyzed as treated). Of the 420 subjects randomized, 418 instilled at least one dose of study medication and were included in the safety population; one subject randomized to BOL-303259-X received timolol in the efficacy phase and was therefore analyzed as part of the timolol treatment group.
Measure: Count of Participants; unit: Participants
Groups:
- BOL-303259-X: BOL-303259-X ophthalmic solution QD (PM) and vehicle QD (AM) administered for 3 months into the study eye during the efficacy phase.
- Timolol: Timolol maleate ophthalmic solution, 0.5%, administered BID for 3 months into study eye during the efficacy phase.
- BOL-303259-X Safety Extension Phase: Following completion of the efficacy phase, all subjects were converted to BOL-303259-X ophthalmic solution QD (PM) and vehicle QD (AM) for an additional 9 months from Visit 6 through Visit 9 (1 year) during the open label safety extension phase
Arm/Group | BOL-303259-X | Timolol | BOL-303259-X Safety Extension Phase
Number analyzed (Participants) | 283 | 135 | 385
Participants
  >/= 1 nonocular AE | 36 | 19 | 62
  >/= 1 ocular (Study eye) AE | 38 | 16 | 46
Statistical Analysis 1: Comparison: BOL-303259-X vs Timolol; Test type: Other; No statistical analysis was performed on these proportions

ADVERSE EVENTS:
Time Frame: 1 year
Description: Safety Population (analyzed as treated). Of 420 subjects randomized, 418 instilled >/=1 dose and were included in the Safety Population; 1 subject randomized to BOL-303259-X received timolol and was therefore analyzed as part of the timolol group in the efficacy phase of the study. All subjects were converted to BOL-303259-X during the safety extension phase and AEs reported during that phase are presented below as a third arm
Arm/Group | BOL-303259-X | Timolol | BOL-303259-X Safety Extension Phase
Serious Adverse Events (participants affected / at risk) | 3/283 | 2/135 | 8/385
Other Adverse Events (participants affected / at risk) | 11/283 | 3/135 | 5/385
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BOL-303259-X (N=283) | Timolol (N=135) | BOL-303259-X Safety Extension Phase (N=385)
torn rotator cuff (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spider bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Recurrence of breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Allergic angioedema due to Motrin (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Leg disco-ordination (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Right upper lobe lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Fracture of right femoral neck (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dislocation of intraocular lens (General disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BOL-303259-X (N=283) | Timolol (N=135) | BOL-303259-X Safety Extension Phase (N=385)
Eye irritation (Eye disorders) | 11 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No